CLINICAL TRIAL: NCT00469430
Title: Randomized Study of Conservative Versus Surgical Treatment of Appendicitis; Analyses of Result and Economics
Brief Title: Study of Conservative Versus Surgical Treatment of Appendicitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Jeanette Hansson, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-Hansson
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Appendicitis
Keywords: appendicitis; treatment; antibiotics
MeSH Terms: conditions — Appendicitis | interventions — Cefotaxime; Benchmarking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Op (No Intervention): traditional surgery
- Ab (Experimental): antibiotic treatment
  Interventions: Drug: cefotaxim and metronidazol

INTERVENTIONS:
Drug: cefotaxim and metronidazol — iv administration for at least 24 h
  Arms: Ab

SUMMARY:
The purpose of this study is to determine if antibiotic treatment of appendicitis is an option compared to surgery. The investigators' hypothesis is that a majority of patients with appendicitis can heal without surgery and that there are several advantages with antibiotic treatment related to time to recover, complications and economical aspects.

DETAILED DESCRIPTION:
Appendicitis is a common disease; 1/1000 gets it every year. 7% will get appendicitis during their lifetime. Surgery, open or laparoscopic, is the traditional treatment. A number of these patients don´t have appendicitis when operated on and the operation is therefore unnecessarily performed. It is also a risk for complications after surgery; for instance wound infection, postoperative small bowel obstruction.

In our study we will compare antibiotic as the only treatment with traditional surgical treatment. Patients with "suspected appendicitis" are randomized to either surgery or antibiotics according to their birth date.

Patients in "the surgery group" are treated according to standard routines. Patients in "the antibiotic group" are treated with intravenous antibiotics for at least 24h - this regime can be prolonged if clinical recovery doesn´t occur - and submitted from hospital with oral antibiotics. If patients in the antibiotic group deteriorate during the hospital stay (suspicious perforation) they will be operated.

Parameters that will be analyzed are:

* primary healing in the antibiotic group
* frequency of relapse in appendicitis in the antibiotic group
* complications in both groups
* economical analysis (hospital stay, sick leave time, time off work) in both groups

ELIGIBILITY:
Inclusion Criteria:

* Suspected appendicitis in patients over 18 years

Exclusion Criteria:

* Under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2006-05; Primary Completion 2007-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
treatment efficacy | one year

SECONDARY OUTCOMES:
complications | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kent Lundholm, Principal Investigator — Göteborg University
Locations (1):
- Göteborg University, Sahlgrenska Universitetssjukhuset, Gothenburg, Göteborg, Sweden

REFERENCES:
- [Background] Eriksson S, Granstrom L. Randomized controlled trial of appendicectomy versus antibiotic therapy for acute appendicitis. Br J Surg. 1995 Feb;82(2):166-9. doi: 10.1002/bjs.1800820207. PMID 7749676
- [Background] Styrud J, Eriksson S, Nilsson I, Ahlberg G, Haapaniemi S, Neovius G, Rex L, Badume I, Granstrom L. Appendectomy versus antibiotic treatment in acute appendicitis. a prospective multicenter randomized controlled trial. World J Surg. 2006 Jun;30(6):1033-7. doi: 10.1007/s00268-005-0304-6. PMID 16736333
- [Derived] Hansson J, Korner U, Khorram-Manesh A, Solberg A, Lundholm K. Randomized clinical trial of antibiotic therapy versus appendicectomy as primary treatment of acute appendicitis in unselected patients. Br J Surg. 2009 May;96(5):473-81. doi: 10.1002/bjs.6482. PMID 19358184